CLINICAL TRIAL: NCT00644605
Title: A Multinational, Multi-centre, Randomised, Double-blind, Double-dummy, Placebo-controlled Study to Assess the Efficacy and Safety of 20, 40, and 80mg TID Sildenafil in the Treatment of Pulmonary Arterial Hypertension in Subjects Aged 18 Years and Over
Brief Title: A Study to Assess the Efficacy and Safety of 20, 40, and 80mg of Sildenafil Three Times a Day in the Treatment of Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481140
Record Dates: First submitted 2008-03-20; First posted 2008-03-27 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Active Comparator)
  Interventions: Drug: sildenafil
- Arm 2 (Active Comparator)
  Interventions: Drug: sildenafil
- Arm 3 (Active Comparator)
  Interventions: Drug: sildenafil
- Arm 4 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sildenafil — sildenafil 40 mg by mouth three times daily (TID), with doses at least 6 hours apart, for 12 weeks
  Arms: Arm 2
Drug: sildenafil — sildenafil 80 mg by mouth three times daily (TID), with doses at least 6 hours apart, for 12 weeks; initially, patients received 40mg TID for one week and were then up-titrated to 80mg TID
  Arms: Arm 3
Drug: placebo — placebo by mouth three times daily (TID), with doses at least 6 hours apart, for 12 weeks
  Arms: Arm 4
Drug: sildenafil — sildenafil 20 mg by mouth three times daily (TID), with doses at least 6 hours apart, for 12 weeks
  Arms: Arm 1

SUMMARY:
To evaluate the effect of three doses of oral sildenafil (20, 40 and 80 mg three times a day [TID]) on exercise capacity, as measured by the 6-Minute Walk test, as well as the safety and tolerability, after 12 weeks of treatment in subjects with pulmonary arterial hypertension who are aged 18 years and over. To investigate the plasma concentration-effect relationship and to determine the population pharmacokinetic (PK) parameters.

ELIGIBILITY:
Inclusion Criteria:

Included patients had primary pulmonary arterial hypertension, pulmonary hypertension secondary to connective tissue disease, or pulmonary hypertension with surgical repair at least 5 years previously; a mean pulmonary artery pressure greater than or equal to 25 mmHg and a pulmonary artery wedge pressure of less than or equal to 15 mmHg at rest, via right heart catheterisation within 21 days prior to randomisation; and a baseline 6-Minute Walk test distance of 100 m to 450 m.

Exclusion Criteria:

Subjects with congenital heart disease, pulmonary hypertension due to thromboembolism, HIV, chronic obstructive airway disease, congestive heart failure or schistosomiasis; subjects with significant (ie > 2+) valvular disease other than tricuspid regurgitation or pulmonary regurgitation; and acutely decompensated heart failure within the previous 30 days; subjects with pulmonary hypertension secondary to any other etiology other than those specified in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2002-10; Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in exercise capacity, as measured by distance walked in six minutes (6-Minute Walk test). | Week 12

SECONDARY OUTCOMES:
Change from baseline in mean pulmonary arterial pressure | Week 12
Time from randomisation to the first occurrence of clinical worsening (death or lung transplantation or hospitalisation due to pulmonary hypertension or initiation of prostacyclin therapy or initiation of bosentan therapy) | Week 0 to 12
Change from baseline in the BORG dyspnoea score | Week 12
Change from baseline in pulmonary hypertension criteria for functional capacity and therapeutic class | Week 12
Change from baseline in the 8 dimensions of SF-36 (Physical functioning, Role functioning, Bodily pain, General health, Vitality, Social functioning, Mental health and Reported health transition) | Week 4 and Week 12
Change from baseline at Weeks 4 and 12 in the 5 dimensions of ED5Q (Mobility, Self care, Usual Activities, Pain/Discomfort and Anxiety/Depression) | Week 4 and Week 12
Patient overall preference assessment | Week 12
Change in Chronic Use of Background Therapy for Pulmonary Arterial Hypertension | throughout the study
Change from baseline in hemodynamic parameters | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (57):
- United States (18):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Australia (2):
  - Pfizer Investigational Site, Darlinghurst, New South Wales
  - Pfizer Investigational Site, Melbourne, Victoria
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Leuven
- Pfizer Investigational Site, São Paulo, São Paulo, Brazil
- Pfizer Investigational Site, Prague, Czechia
- Pfizer Investigational Site, Copenhagen, Denmark
- Pfizer Investigational Site, Clamart, France
- Germany (4):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Giessen
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, Leipzig
- Pfizer Investigational Site, Shatin N T, Hong Kong
- Hungary (2):
  - Pfizer Investigational Site, Budapest, Pest County
  - Pfizer Investigational Site, Zalaegerszeg, Zala County
- Israel (2):
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Tel Litwinsky
- Italy (2):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Pisa
- Pfizer Investigational Site, Kuala Lumpur, Malaysia
- Pfizer Investigational Site, Tlalpan, Mexico
- Pfizer Investigational Site, Amsterdam, Netherlands
- Pfizer Investigational Site, Oslo, Norway
- Poland (3):
  - Pfizer Investigational Site, Katowice
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Zabrze
- Pfizer Investigational Site, Singapore, Singapore
- South Africa (3):
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Johannesburg
  - Pfizer Investigational Site, Parow
- Pfizer Investigational Site, Suwon, South Korea
- Spain (2):
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
- Sweden (2):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Mölndal
- United Kingdom (4):
  - Pfizer Investigational Site, Papworth Everard, Cambridgeshire
  - Pfizer Investigational Site, Sheffield, South Yorkshire
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, HIGH Heaton, Newcastle-upon-tyne

REFERENCES:
- [Derived] Wirostko BM, Tressler C, Hwang LJ, Burgess G, Laties AM. Ocular safety of sildenafil citrate when administered chronically for pulmonary arterial hypertension: results from phase III, randomised, double masked, placebo controlled trial and open label extension. BMJ. 2012 Feb 21;344:e554. doi: 10.1136/bmj.e554. PMID 22354598
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481140&StudyName=A%20multinational%2C%20multi-center%2C%20randomized%2C%20double-blind%2C%20double-dummy%2C%20placebo-controlled%20study%20to%20assess%20the%20efficacy%20and%20safety%20of%202